CLINICAL TRIAL: NCT07382544
Title: Phase 1b Trial of Combined PRMT5 Inhibition With BMS-986504 and PARP Inhibition With Olaparib in Patients With Advanced Cancer With MTAP Loss
Brief Title: Phase 1b Trial of BMS-986504 in Combination With Olaparib in Patients With MTAP Loss
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-1200; NCI-2025-09342 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2025-12-29; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Advanced Cancer; Solid Tumor
MeSH Terms: interventions — olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Part A Dose Escalation: Treatment with BMS-986504 + Olaparib (Experimental): Study treatment will be administered on an outpatient basis
  Interventions: Drug: MRTX1719; Drug: Olaparib
- Part B Pharmacodynamic Expansion Cohort 1: Treatment with BMS-986504 at C1D1 + Olaparib at C1D15 (Experimental): Study treatment will be administered on an outpatient basis
  Interventions: Drug: MRTX1719; Drug: Olaparib
- Part B Pharmacodynamic Expansion Cohort 2: Treatment with Olaparib at C1D1 + BMS-986504 at C1D15 (Experimental): Study treatment will be administered on an outpatient basis
  Interventions: Drug: MRTX1719; Drug: Olaparib

INTERVENTIONS:
Drug: MRTX1719 — Given by mouth
Drug: Olaparib — Given by mouth
  Other Names: Lynparza

SUMMARY:
The goal of this clinical research study is to learn about the safety and effects of BMS-986504 in combination with olaparib in patients with advanced solid tumors with MTAP loss.

DETAILED DESCRIPTION:
Primary Objective:

1. To determine the safety and tolerability of BMS-986504 in combination with olaparib in patients with advanced solid tumors with MTAP loss.

Secondary Objectives:

1. To characterize the PK profile of BMS-986504 in combination with olaparib in patients with advanced solid tumors with MTAP loss.
2. To determine the preliminary antitumor activity of BMS-986504 in combination with olaparib with advanced solid tumors with MTAP loss.
3. To evaluate the pharmacodynamic activity of BMS-986504 in combination with olaparib in advanced solid tumors with MTAP loss.
4. To evaluate predictors of response and resistance to BMS-986504 in combination with olaparib in patients with advanced solid tumors with MTAP loss.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years.
2. All patients must have a histologically confirmed advanced or metastatic solid tumor that has been refractory to standard therapy or are not eligible for standard therapy and have no alternative curative-intent treatment options at the time of patient enrollment. For the dose escalation, any solid tumor is eligible, but enrollment will be enriched for CCA and pancreatic cancer. For the pharmacodynamic expansion, patients must have histologically confirmed advanced or metastatic CCA or pancreatic cancer.
3. Homozygous deletion of MTAP as detected by Clinical Laboratory Improvement Amendmentscertified next-generation sequencing test or absence of MTAP protein as detected by CLIAcertified immunohistochemistry test.
4. Patients in Part A must have archived tumor tissue available for retrospective analysis or agree to pre-treatment biopsy.
5. Ability to understand and the willingness to sign a written informed consent document.
6. Ability to comply with the study protocol, in the investigator's judgment.
7. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 (Appendix 1).
8. Life expectancy ≥3 months.
9. Patients in the pharmacodynamic expansion must have measurable and biopsiable disease per the RECIST v1.1 (Appendix 2). Patients in the dose escalation can have evaluable or measurable disease.
10. Patients must have adequate washout from prior therapy at the time of study treatment initiation: 3 weeks from any treatment specifically for systemic tumor control: 5 half-lives from small molecule targeted agents and ≥ 2 weeks from radiotherapy (except for patients with brain metastasis treatment with Gamma Knife; in these cases, > 1 week is required). Palliative radiotherapy is permitted for a preexisting lesion, provided it does not interfere with the assessment of tumor target lesions (e.g., the lesion to be irradiated must not be a site of measurable disease).
11. Patients must have recovered from toxicities of prior anticancer therapy (Grade ≤ 1 toxicity) except for alopecia and peripheral neuropathy.
12. Adequate organ and marrow function as defined below within 28 days prior to study treatment initiation:

    * Hemoglobin ≥ 9.0 g/dL
    * Absolute neutrophil count (ANC) ≥ 1500/mm3
    * Platelets ≥ 100,000/mm3
    * Adequate renal function: Estimated glomerular filtration rate ≥ 50 mL/min/1.73 m2 by the Chronic Disease Epidemiology Collaboration equation; estimated creatinine clearance ≥50 mL/min (calculated using institutional standard method).
    * Adequate hepatic function: Total bilirubin ≤ 1.5 × upper limit of normal (ULN); Patients with Gilbert's syndrome with total bilirubin ≤ 2.0 × ULN and direct bilirubin within normal limits are permitted; Aspartate aminotransferase/ALT ≤ 3 × institutional ULN or ≤ 5 × ULN for patients with liver metastases.
    * For patients not receiving therapeutic anticoagulation: international normalized ratio or activated partial thromboplastin time ≤1.5 × ULN. For patients receiving therapeutic anticoagulation: stable anticoagulant regimen.
13. Patients must be able to take PO medications.
14. Women of childbearing potential (WOCBP) must have a negative serum pregnancy test result within 72 hours prior to study treatment initiation.

WOCBP must agree to use adequate contraception as described below from the screening visit through at least 6 months after the last dose of study treatment. (Refer to Pregnancy Assessment Policy MD Anderson Cancer Center [MDACC] Institutional Policy # CLN1114). This includes all female patients, between the onset of menses (as early as 8 years of age) and 55 years unless the patient presents with an applicable exclusionary factor which may be one of the following:

* Postmenopausal (no menses in ≥ 12 consecutive months).
* History of hysterectomy or bilateral salpingo-oophorectomy.
* Ovarian failure (follicle-stimulating hormone and estradiol in menopausal range and have received whole pelvic radiation therapy).
* History of bilateral tubal ligation or another surgical sterilization procedure.

WOCBP must agree to use a combination of a hormonal and a non-hormonal contraceptive method or a non-hormonal method alone that is highly effective (with a failure rate of < 1% per year: copper intrauterine device) during the intervention period and for at least 6 months after the last dose of study intervention, or according to approved local product label requirements for individual chemotherapy agents, whichever is longer.

WOCBP are not permitted to use hormonal contraceptive methods alone as a highly effective method of contraception and must use an additional non-hormonal highly effective method of contraception.

WOCBP must also agree not to donate eggs (ova, oocytes) for the purpose of reproduction for the same period. Participants should be advised to seek advice about egg donation and cryopreservation of germ cells before treatment.

Exclusion Criteria:

1. Part B only: Prior treatment with a PRMT5 or methionine adenosyltransferase 2A inhibitor.
2. Patients who have a known additional malignancy that is progressing or requires active treatment at time of study treatment initiation. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin that has undergone potentially curative therapy, and in situ cervical cancer.
3. Patients with meningeal carcinomatosis, leptomeningeal carcinomatosis, spinal cord compression, or symptomatic or unstable brain metastases. Note: Patients with stable brain metastases (defined as asymptomatic or no requirement for high-dose or increasing dose of systemic corticosteroids and without imminent need of radiation therapy) are eligible (including those with untreated brain metastases). If applicable, patients must have completed brain radiation therapy and recovered adequately from any associated toxicity and/or complications prior to eligibility assessment.
4. Concomitant use of strong cytochrome P450 (CYP)3A inhibitors or inducers are prohibited within 14 days or 5 half-lives, whichever is longer, prior to study treatment initiation and during the study treatment period. For a comprehensive list of CYP3A inhibitors/inducers, refer to: https://www.fda.gov/drugs/drug-interactions-labeling/drug-development-and-drug-interactionstable-substrates-inhibitors-and-inducers.
5. Any clinically significant comorbidities such as uncontrolled pulmonary disease, known impaired cardiac function or clinically significant cardiac disease (including but not limited to known left ventricular ejection fraction < 50%, congenital long QT syndrome, corrected QT interval using Fridericia's formula ≥ 480 msec on screening electrocardiogram [ECG], unstable angina pectoris ≤ 3 months prior to study treatment initiation, and acute myocardial infarction ≤ 3 months prior to study treatment initiation), or any other condition that could compromise the patient's participation in the study.
6. Treatment with a live, attenuated vaccine within 4 weeks prior to study treatment initiation.

   Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster, yellow fever, rabies, Bacille Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., FluMist®) are live attenuated vaccines and are not allowed. Non-live COVID vaccines will be allowed on study, but it is recommended to avoid their use during the first treatment cycle (from 3 days prior to Cycle 1 Day 1 through Cycle 2 Day 3).
7. Concomitant use of medications known to be sensitive substrates of breast cancer resistance protein (including, but not limited to, rosuvastatin and sulfasalazine) or P-glycoprotein (P-gp; including, but not limited to, dabigatran etexilate, digoxin, fexofenadine).
8. Patients who are pregnant or breastfeeding or expecting to conceive within the projected duration of the study, starting with the screening visit through 7 months after the last dose of study treatment.
9. Any known psychiatric, substance abuse, or other disorder that would interfere with cooperation with the requirements of the study, in the opinion of the investigator.
10. Patients who are receiving any other investigational agents.
11. History of allergic reactions attributed to compounds of similar chemical or biologic composition to the study drugs.
12. Patients who have an active infection requiring intravenous (IV) antibiotics.
13. Patients with any gastrointestinal disorder that would significantly alter the absorption of the study drugs (e.g., active ulcerative diseases, uncontrolled nausea, uncontrolled vomiting, uncontrolled diarrhea, malabsorption syndrome).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2030-01-31 (Estimated); Study Completion 2032-01-31 (Estimated)

PRIMARY OUTCOMES:
Safety and Adverse Events (AEs) | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Jordi Rodon Ahnert, MD, PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- The University of Texas M. D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org